CLINICAL TRIAL: NCT00764101
Title: Effects of Attentional Bias Modification on Attentional Bias and Symptoms of Posttraumatic Stress Disorder
Brief Title: Attentional Bias Modification in Patients With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PsyQ (Other)
Collaborators: Leiden University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Willem Van der Does, PhD, Leiden University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60-60105-98-128
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 9 sessions of attentional bias modification (computerized training program)
  Interventions: Behavioral: Attentional Bias Modification
- 2 (Placebo Comparator): Attentional control condition (placebo training program)
  Interventions: Behavioral: Attentional Bias Modification

INTERVENTIONS:
Behavioral: Attentional Bias Modification — computerized training to reduce attentional bias in posttraumatic stress disorder
  Other Names: Attentional Training

SUMMARY:
Randomized, placebo-controlled trial of 9 sessions of computerized attentional bias training on attentional bias and on symptoms of Posttraumatic Stress Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Posttraumatic Stress Disorder

Exclusion Criteria:

* Diagnosis of psychosis, drug- or alcohol dependency/abuse;
* Unable to fill in questionnaires in Dutch;
* Color blindness (Stroop test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | End of Trial + 3 week Follow-Up

SECONDARY OUTCOMES:
PTSD symptoms (self-report) | end of trial + 3wk Follow Up
Attentional Bias (dot-probe test) | End of trial + 3wk Follow-up
Emotional Stroop Interference | End of trial + 3wk Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Willem van der Does, professor, Study Director — Leiden University; Maartje Schoorl, MS, Principal Investigator — PsyQ Nederland bv
Locations (1):
- PsyQ Haaglanden, department of psychotrauma, The Hague, South Holland, Netherlands

REFERENCES:
- [Derived] Schoorl M, Putman P, Van Der Does W. Attentional bias modification in posttraumatic stress disorder: a randomized controlled trial. Psychother Psychosom. 2013;82(2):99-105. doi: 10.1159/000341920. Epub 2012 Dec 22. PMID 23295710